CLINICAL TRIAL: NCT06680817
Title: Real-World, Long-Term Data Collection to Gain Clinical Insights Into Faricimab (FaReal Study)
Brief Title: A Real-World Study to Gain Clinical Insights Into Faricimab (FaReal Study)
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MR45586
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Faricimab for nAMD: This cohort will be divided into two sub-cohorts based on eye treatment history: anti-VEGF treatment naive and anti-VEGF pre-treated.
  Interventions: Drug: Faricimab
- Cohort 2: Faricimab for DME: This cohort will be divided into two sub-cohorts based on eye treatment history: anti-VEGF treatment naive and anti-VEGF pre-treated.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered as per local clinical practice and local labeling.
  Other Names: VABYSMO®; RO6867461; RG7716

SUMMARY:
The FaReal study aims to evaluate the effectiveness, safety, clinical insights and treatment patterns in patients treated with faricimab, in neovascular age-related macular degeneration (nAMD) or diabetic macular edema (DME) in at least one eye, in real-world routine clinical practice over a 2-year patient follow-up period. Additionally, the FaReal study also aims to describe and evaluate health economic aspects of previous anti-VEGF treatments and current treatment with faricimab.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving faricimab according to the local faricimab product label and who have initiated treatment with faricimab at time of the ICF signature date or no more than 3 months prior to the ICF signature date, in diabetic macular edema (DME) or neovascular age-related macular degeneration (nAMD) in at least one eye
* Patients have received at least one faricimab treatment (the first dose) in the study eye
* Patients should have available data for visual acuity (VA) and Central Subfield Thickness (CST) for the Baseline level (i.e. examinations to be performed at the index date or within 4 months prior to it)

Exclusion Criteria:

* Patient participation in any investigational ophthalmology clinical trial that includes receipt of any ophthalmological investigational drug or procedure within the last 28 days prior to the ICF signature date
* Concomitant participation in any interventional clinical study
* Active ocular inflammation and/or suspected/active ocular infection in either eye
* Patients treated with faricimab who have and are currently participating in patient support programs (PSP) that are Market Research and Patient Support Programs (MAP) including Post Trial Access Programs (PTAP) and Compassionate Use Programs (CUP)
* Patients with non-ocular sight threatening disease which have an effect on the primary endpoint (e.g., apoplexia)
* Hypersensitivity to the active substance or any of the excipients of Vabysmo (as per label)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated with faricimab approved for nAMD and DME in real-world, routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Acuity from Index Date to 12 Months | Index Date and 12 months
  The index date is defined as the date of the first faricimab treatment injection in the eye.

SECONDARY OUTCOMES:
Change in Visual Acuity from Index Date to 3, 6, and 24 Months | Index Date and 3, 6, and 24 months
Change in Central Subfield Thickness (CST) from Index Date to 3, 6, 12, and 24 Months | Index Date and 3, 6, 12, and 24 months
Percentage of Eyes on Each Treatment Regimen (Fixed, Treat-and-Extend, As Needed, or Other) Over Time | Index Date and 3, 6, 12, and 24 months
Number of Faricimab Intravitreal Injections per Eye per Year | 12 and 24 months
Number of Faricimab Intravitreal Injections in the Loading Phase for Participants who are anti-VEGF Treatment Naive or anti-VEGF pre-Treated | Approximately 4 months
Total Number of Visits and Number of Visits With or Without Treatment Over Time | 3, 6, 12, and 24 months
Cumulative Time Spent in Each Treatment Regimen (Fixed, Treat-and-Extend, As Needed, or Other) | From Index Date to 24 months
Percentage of Eyes With Treatment Switch from Faricimab by Reason for Switch in Participants who are anti-VEGF Treatment Naive or anti-VEGF pre-Treated | 3, 6, 12, and 24 months
Percentage of Eyes Obtaining Treatment Intervals of Once Every 8, 12, or 16 Weeks or Other Intervals in Participants who are anti-VEGF Treatment Naive or anti-VEGF pre-Treated | 12 and 24 months
Change in Visual Acuity from Index Date Over Time, According to Treatment Regimen (Fixed, Treat-and-Extend, As Needed, or Other) | Index Date and 3, 6, 12, and 24 months
Change in Visual Acuity from Index Date Over Time, According to Number of Intravitreal Treatments | Index Date and 3, 6, 12, and 24 months
Change in Visual Acuity from Index Date Over Time, According to Total Number of Visits | Index Date and 3, 6, 12, and 24 months
Change in Visual Acuity from Index Date Over Time, According to Treatment Intervals | Index Date and 3, 6, 12, and 24 months
Change in Visual Acuity from Index Date Over Time, According to Type of anti-VEGF Pre-Treatment and Number of Previous Injections for Preceding Regimen at Index Date | Index Date and 3, 6, 12, and 24 months
Change in Visual Acuity from Index Date Over Time, According to Length of Diagnosis of Disease at Index Date | Index Date and 3, 6, 12, and 24 months
Number of Participants with at Least One Ocular Adverse Event | Approximately 2 years
Number of Participants with at Least One Non-Ocular Adverse Event | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- Austria (5):
  - LKH-Univ.Klinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Kepler Universitätskliniken GmbH - Med Campus III, Linz
  - Medizinische Universitat Wien, Vienna
  - Hanusch Krankenhaus, Vienna
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment Trimontium OOD Plovdiv;Ophthalmology, Plovdiv
  - Eye Medical Center St. Luka, Plovdiv
  - Eye Diseases Medical Center LUX OPTICS;ophthalmology, Sofia
  - Tokuda Hospital, Sofia
  - Medical Clinic Svetlina, Sofia
  - Ambulatory for Group Practice for Specialized Medical Care in Ophthalmology - Dr. Grupchevi OOD;Ophthalmology, Varna
- Czechia (5):
  - Krajska nemocnice Liberec a.s., Liberec
  - Klaudianova Nemocnice - Mlada Boleslav;Ophtalmology dpt, Mladá Boleslav
  - Fakultni nemocnice Olomouc, Olomouc
  - Faculty Hospital Ostrava, Ostrava
  - Ustredni vojenska nemocnice - Vojenska fakultni nemocnice Praha, Prague
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Greece (4):
  - General Hospital of Athens "Korgialeneio - Benakeio" Hellenic Red Cross, Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Larissa, Larissa
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Erzsebet Furdo Gyogyaszati es Szurokozpont, Miskolc
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudományegyetem ÁOK, Szeged
- Ireland (2):
  - Mater Private Hospital, Dublin
  - Institute of Eye Surgery, Waterford
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Shamir Medical Center Assaf Harofeh, Beer Jacob
  - Soroka university medical center, Beersheba
  - Carmel medical center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Latvia (3):
  - Pauls Stradins Clinical University hospital, Riga
  - Riga East Clinical University hospital Bikernieki, Riga
  - Latvian-American Eye Center, Riga
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - ETZ Elisabeth, Tilburg
- Poland (7):
  - NZOZ Specjalistyczna Poradnia Lekarska Adrian Wojciech Przystupa, Bielsk Podlaski
  - Centrum Uslug Medycznych OKO-MED, Grudziądz
  - USK Nr 2 im. WAM w Lodzi, Centralny Szpital Weteranow, Lodz
  - Szpital Wojewodzki w Poznaniu, Poznan
  - Pomorski Uniwersytet Medyczny, Szczecin
  - Szpitale Pomorskie, Szpital Specjalistyczny im. F. Ceynowy, Wejherowo
  - Szpital Uniwersytecki im. Karola Marcinkowskiego w Zielonej Górze, Zielona Góra
- Portugal (5):
  - Espaco Medico Coimbra, Coimbra
  - ULS Lisboa Ocidental - Hospital Egas Moniz, Lisbon
  - Hospital CUF Tejo, Lisbon
  - IMO - Instituto de Microcirurgia Ocular, Lisbon
  - Hospital de Sao Joao, Porto
- Slovakia (4):
  - Nemocnica s poliklinikou Trebišov, a.s., Trebišov
  - Fakultna nemocnica Trencin Ocna klinika, Trenčín
  - Fakultna nemocnica Trnava, Trnava
  - OFTAL s.r.o. Specializovana nemocnica v odbore oftalmologia Zvolen, Zvolen
- General Hospital Murska Sobota, Murska Sobota, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing